CLINICAL TRIAL: NCT01865838
Title: A Study Into the Effect of Seprafilm on Post Operative Adhesions After Open Total Thyroidectomy.
Brief Title: A Study Into the Effect of Seprafilm in Open Total Thyroidectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: safety issue
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Seprafilm in Thyroidectomy
Record Dates: First submitted 2013-05-14; First posted 2013-05-31 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Thyroid Carcinoma
Keywords: Total thyroidectomy; Seprafilm; Swallowing difficulty post thyroidectomy
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Seprafilm (Sanofi, USA) (Active Comparator): Patients in this arm received Seprafilm during surgery.
  Interventions: Device: Seprafilm (Sanofi, USA)
- Control (No Intervention): Patients in this arm does NOT receive Seprafilm during surgery.

INTERVENTIONS:
Device: Seprafilm (Sanofi, USA) — Studies have unequivocally shown that Seprafilm is effective in reducing internal adhesion formation after abdominal surgery. In a large scaled randomized controlled trial involving about 1700 patients, Fazio et al. found that the use or Seprafilm reduces the risk of small bowel intestinal obstruction which required operative intervention. The safety profile of Seprafilm has also been nicely demonstrated in a randomized controlled trial by Beck et al. in this study, the authors concluded that within the context of abdomino-pelvic surgery, Seprafilm does not increase the incidence of abdominal/pelvic abscesses in patients after abdomino-pelvic surgery; if anything, the anti-adhesive properties of Seprafilm are such that the authors noted an increased risk of anastomotic complications in patients whose bowel anastomoses were in close contact with Seprafilm.
  Arms: Seprafilm (Sanofi, USA)

SUMMARY:
The investigators intend to determine the role of Seprafilm, a popular anti-adhesive agent in minimising internal adhesion formation in the neck after thyroid surgery and therefore reduce swallowing discomfort experienced by patients after surgery.

DETAILED DESCRIPTION:
Thyroid surgery not only constitutes one of the main pillars in the treatment of thyroid cancers, but is also employed in the management of symptomatic goitres. Occasionally, it is mandated in patients with thyrotoxicosis refractory to medical therapy. While thyroid surgery can be performed with low risks such that patients rarely have to stay beyond three days in hospital, the track record of thyroid surgery is somewhat blemished by the unfortunate side effects associated with the neck scarring after thyroid surgery. Not uncommonly, patients experience discomfort in the neck region after thyroid surgery; in the extreme of cases, patients may even complain of a lifelong pulling sensation in the neck area during eating.

The anti-adhesive properties of Seprafilm are well established in animal studies and affirmed by clinical observations in abdominal surgeries that utilize this material. Thus, Seprafilm is routinely used in instances when a surgeon foresees a need to perform abdominal surgery on the same patient in future, or during the fashioning of a temporary stoma. The safety profile of Seprafilm in thyroidectomy has also been shown by a recent study conducted by a group of clinicians in Seoul.

We postulate that the application of Seprafilm to the surgical wound towards the end of a thyroidectomy significantly reduces internal adhesion formation in the neck region. By achieving this objective, we hope to improve patients' satisfaction with thyroid surgery in terms of ease of swallowing after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-75
* Histological confirmation of differentiated thyroid cancer requiring surgery, symptomatic goiters, thyroid nodules requiring histological analysis, or thyrotoxicosis poorly controlled by medication.
* Undergoing total thyroidectomy

Exclusion Criteria:

* Previous neck surgery
* Previous neck radiotherapy
* Patients with a known history of keloids
* Patients with a known history of motility disorders in the upper gastrointestinal tract and preexisting swallowing difficulty.
* Patients with metastatic disease; patients with disease that would require postop radiation therapy, radionuclide iodine therapy and any adjuvant therapies.
* Patients with advanced disease that would require radical or modified neck dissection
* Patients with lobe larger than 10 cm, or nodule larger than 8 cm which require extensive dissection that may confound the study
* Patients with connective tissue diseases and chronic diseases on long-term medications that may interfere with wound healings such as steroids

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Cricoid elevation | 1 to 14 days before the surgery, postop day 14 and 3 months postop
  Trial candidates are to undergo videofluoroscopy to assess their swallowing and cricoid elevation is measured using ImageJ.
  * First measurement is 1 to 14 days before the surgery.
  * Second measurement is 14 days postop.
  * Third measurement is 3 months postop.

SECONDARY OUTCOMES:
Hyoid elevation | 1 to 14 days before the surgery, postop day 14 and 3 months postop
  Trial candidates are to undergo videofluoroscopy to assess their swallowing and hyoid elevation is measured using ImageJ.
  * First measurement is 1 to 14 days before the surgery.
  * Second measurement is 14 days postop.
  * Third measurement is 3 months postop.
Crico-hyoid distance | 1 to 14 days before the surgery, postop day 14 and 3 months postop
  Trial candidates are to undergo videofluoroscopy to assess their swallowing and hyoid elevation is measured using ImageJ.
  * 1 to 14 days before the surgery
  * Second measurement is 14 days postop.
  * Third measurement is 3 months postop.
Videotaping measurement | 1 to 14 days before the surgery, postop day 14 and 3 months postop
  Trial candidates are to undergo videotaping of their surgical incision site during swallowing. Maximal displacement of the incision site will be measured and recorded using ImageJ.
  * First measurement is 1 to 14 days before the surgery.
  * Second measurement is 14 days postop.
  * Third measurement is 3 months postop.
Swallowing Quality of Life questionaire | 1 to 14 days before the surgery, postop day 14 and 3 months postop
  Trial candidates will be interviewed regarding their swallowing using the Sydney Swallowing questionnaire. Patients will be interviewed three times.
  * First interview is 1 to 14 days before the surgery.
  * Second interview is 14 days postop.
  * Third interview is 3 months postop.

OTHER OUTCOMES:
Duration of surgery | During surgery
  -Knife-to-skin time to closure.
Drainage | Day 1 to Day 3 after the surgery
  -Surgical drain will be placed for patients at surgeons' discretion. Drain amount will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Khoon H Tan, MBBS, PhD, Principal Investigator — National Cancer Centre, Singapore
Locations (2):
- Singapore (2):
  - Singapore General Hospital, Singapore
  - National Cancer Centre Singapore, Singapore

REFERENCES:
- [Background] Fazio VW, Cohen Z, Fleshman JW, van Goor H, Bauer JJ, Wolff BG, Corman M, Beart RW Jr, Wexner SD, Becker JM, Monson JR, Kaufman HS, Beck DE, Bailey HR, Ludwig KA, Stamos MJ, Darzi A, Bleday R, Dorazio R, Madoff RD, Smith LE, Gearhart S, Lillemoe K, Gohl J. Reduction in adhesive small-bowel obstruction by Seprafilm adhesion barrier after intestinal resection. Dis Colon Rectum. 2006 Jan;49(1):1-11. doi: 10.1007/s10350-005-0268-5. PMID 16320005
- [Background] Beck DE, Cohen Z, Fleshman JW, Kaufman HS, van Goor H, Wolff BG; Adhesion Study Group Steering Committee. A prospective, randomized, multicenter, controlled study of the safety of Seprafilm adhesion barrier in abdominopelvic surgery of the intestine. Dis Colon Rectum. 2003 Oct;46(10):1310-9. doi: 10.1007/s10350-004-6739-2. PMID 14530667
- [Background] Park WS, Chung YS, Lee KE, Kim HY, Choe JH, Koh SH, Youn YK. Anti-adhesive effect and safety of sodium hyaluronate and sodium carboxymethyl cellulose solution in thyroid surgery. Asian J Surg. 2010 Jan;33(1):25-30. doi: 10.1016/S1015-9584(10)60005-X. PMID 20497879
- [Background] Metwally M, Cheong Y, Li TC. A review of techniques for adhesion prevention after gynaecological surgery. Curr Opin Obstet Gynecol. 2008 Aug;20(4):345-52. doi: 10.1097/GCO.0b013e3283073a6c. PMID 18660685